CLINICAL TRIAL: NCT06500039
Title: The Effect of Positive Psychological Interventions on Quality of Life and Well-Being in Patients With Multiple Sclerosis
Brief Title: Positive Psychological Interventions for Patients With Multiple Sclerosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Aliye Yaşayacak, Lecturer, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AbantIBU-SBF-AY-01
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis, Quality of Life, Well-Being
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The research was planned as a randomized controlled prospective study. It will be carried out in two groups.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Participants will implement positive psychological interventions at home for four weeks. In the first two weeks, they will do the three good things in life exercise, in the third week, they will write a gratitude letter, and in the fourth week, they will write five things they are grateful for. Participants will be given a guide booklet to write on.
  Interventions: Other: Positive Psychological Intervention Program
- Kontrol group (Placebo Comparator): Control group participants will practice writing their daily routines for four weeks. They will write a few sentences about the nutrition routine in the first week, the hygiene routine in the second week, the sleeping routine in the third week, and the shopping routine in the fourth week. Participants will be given a guide booklet for the writing exercise.
  Interventions: Other: Writing Daily Routines

INTERVENTIONS:
Other: Positive Psychological Intervention Program — An intervention method consisting of three good things in life and gratitude activities was determined for the intervention group. It will take four weeks. Three good deeds will be held for two weeks, and gratitude activities will be held for the last two weeks. Participants will record the interventions on a prepared booklet.
  Arms: Intervention group
Other: Writing Daily Routines — An activity was planned for the control group participants to write their daily routines. They will write down their sleep, nutrition, hygiene and shopping routines, which will be different each week for four weeks. Control group participants will also be given a booklet to write on.
  Arms: Kontrol group

SUMMARY:
This study aims to determine the effectiveness of positive psychological interventions on the quality of life and well-being levels of patients with multiple sclerosis.Two groups will be selected as intervention and control groups. An intervention method consisting of three good things in life and gratitude activities, each lasting two weeks, was determined for the intervention group. An activity was planned for control group participants to write their daily routines.

DETAILED DESCRIPTION:
People with Multiple Sclerosis (MS) face numerous physical and mental symptoms as well as emotional and social challenges. The fact that the disease usually occurs in young adulthood, when individuals are most productive, causes disability, its unpredictable and variable nature, and the lack of a known treatment make it difficult to live with MS and accept the disease. The physical, cognitive, behavioral and social changes that occur with the disease affect daily life activities, well-being. and greatly affects the quality of life. There are various interventions developed to improve the adaptation processes of individuals diagnosed with a chronic disease such as MS, to prevent and reduce psychiatric symptoms, and to increase quality of life and well-being. One of the intervention approaches is positive psychological interventions from the field of positive psychology. Positive psychological interventions are a psychosocial intervention method based on the systematic completion of certain activities aimed at increasing positive emotions, thoughts and behaviors. Since the interventions focus on strengthening positive mental states rather than reducing psychological symptoms, they also have an advantage over traditional interventions in that they can be applied to both sick and non-patients. However, it appears that positive psychological intervention studies have just begun to be implemented in patients with MS. In our country, no study has been found using positive psychological intervention in MS patients. This study aims to determine the effectiveness of positive psychological interventions on the quality of life and well-being levels of patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS by a neurologist according to McDonald criteria
* Having at least 1 year of MS history
* Expanded Disability Status Scale (EDSS) score measured by the neurology clinic is <3.5
* Being between the ages of 18-65 being literate
* Ability to communicate in Turkish
* Volunteering to participate in the study

Exclusion Criteria:

* Having an MS attack and using corticosteroid medication for the last 3 months
* A score of 21 or less on the Montreal Cognitive Assessment (MoCA) test
* Having a mental or organic disability in communicating
* Being diagnosed with any chronic disease other than MS
* Using psychotropic medication or continuing psychotherapy
* Not having or being able to obtain a phone that can connect to the internet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Quality of Life Scale (MSQOL)-54 | six month
  It was developed by Vickrey, Hays, Harooni, Myers, and Ellison (1995). The scale consists of 2 main groups, composite physical health (BFS) and composite mental health (BMS), 12 subgroups and 2 independent items. The reliability coefficients of the scale were found to be between 0.75-0.96, and the test-retest reliability coefficients were found to be between 0.66-0.96. BFS and BMS scores, the two main groups of the MSQOL-54 scale, take a value between 0-100. A high score from the scale indicates a high quality of life.
PERMA Measuring Tool | six month
  It was developed by Butler and Kern (2016) to measure well-being levels. The scale consists of a total of 23 items, 15 items measuring the components of the well-being model and 8 filler items. Among the filler items in the scale, items 7, 12, 14 and 20 are reverse coded. There are 3 items in each dimension of the scale, which consists of 15 items. Sub-dimension scores are calculated by taking the average of the 3 items in the relevant sub-dimension. The Cronbach Alpha internal consistency coefficient for the total score of the scale is 91.

SECONDARY OUTCOMES:
Positive and Negative Mood Scale (PNDS) | six month
  The Positive and Negative Affect Scale was developed by Watson and colleagues (1988) to assess positive and negative emotion. There are a total of 20 items in the scale, 10 items for each subscale. The scale is a five-point Likert scale ranging from 1 (very little to not at all) to 5 (very much). The score a person gets from the positive or negative emotion subscales varies between 10 and 50. The internal consistency coefficients of the original form of the scale are .88 for positive emotion and .85 for negative emotion.

CONTACTS AND LOCATIONS:
Overall Officials: Nazmiye Yıldırım, Study Chair — Bolu Abant İzzet Baysal University; Aliye Yaşayacak, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No